CLINICAL TRIAL: NCT03711721
Title: Nutritional Support to Improve Adherence and Treatment Completion Among HIV-Tuberculosis Co-infected Adults in Senegal, West Africa: A Randomized Pilot Implementation Study
Brief Title: Nutritional Support for HIV-Tuberculosis Co-infected Adults in Senegal, West Africa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: La Clinique des Maladies Infectieuses, Centre Hospitalier National Universitaire de Fann (Unknown)
Responsible Party: Principal Investigator, Noelle Benzekri, Principal Investigator, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 20150056
Record Dates: First submitted 2018-10-08; First posted 2018-10-18 (Actual); Last update posted 2018-10-18 (Actual); Status verified 2018-10

CONDITIONS: HIV and Tuberculosis Co-infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Food basket (Experimental)
  Interventions: Dietary Supplement: Food basket
- Ready-to-Use Therapeutic Food (Experimental)
  Interventions: Dietary Supplement: Ready-to-Use Therapeutic Food

INTERVENTIONS:
Dietary Supplement: Food basket
  Arms: Food basket
Dietary Supplement: Ready-to-Use Therapeutic Food
  Arms: Ready-to-Use Therapeutic Food

SUMMARY:
Food insecurity can contribute to poor adherence to both tuberculosis treatment and antiretroviral therapy (ART). Interventions that target food insecurity have the potential to improve treatment adherence and decrease mortality. The goals of this study were to determine the cost, feasibility, acceptability, and potential impact of implementing nutritional support to improve adherence and treatment completion among HIV-TB co-infected adults in the Casamance region of Senegal, West Africa.

ELIGIBILITY:
Inclusion Criteria:

* HIV-Tuberculosis co-infection
* Age ≥18 years
* Initiating treatment for tuberculosis
* Provide written informed consent

Exclusion Criteria:

• Unwilling or unable to provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Uptake, as determined by percent of monthly nutritional support rations received, transported, stored, and utilized by subjects. | 6 months
Acceptability, as determined by patient reported perceptions of nutritional support. | 6 months
Costs of monthly nutritional support rations. | 6 months

SECONDARY OUTCOMES:
Tuberculosis treatment adherence as determined by Medication Possession Ratio | 6 months
Tuberculosis treatment adherence as determined by patient reported number of missed doses in the previous 7 days and 4 weeks. | 6 months
Tuberculosis treatment completion defined as completing full course of prescribed therapy | 6 months
Adherence to antiretroviral therapy as determined by Medication Possession Ratio | 6 months
Adherence to antiretroviral therapy as determined by patient reported number of missed doses in the previous 7 days and 4 weeks | 6 months
CD4 cell count | 6 months
Presence of acid fast bacteria using sputum smear microscopy | 6 months
Results of GeneXpert | 6 months
Nutritional status as determined by Body Mass Index | 6 months
Nutritional status as determined by change in weight (kg) | 6 months
Food security status measured using the Household Food Insecurity Access Scale (HFIAS) | 6 months
  The HFIAS is a 9-item questionnaire which provides a household food insecurity score on a scale of 1-4, with 1 being not food insecure, 2 being mildly food insecure, 3 being moderately food insecure, and 4 being severely food insecure.
Hemoglobin levels (g/dl) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Noelle A Benzekri, MD, Principal Investigator — University of Washington; Moussa Seydi, MD, Principal Investigator — La Clinique des Maladies Infectieuses, CHNU de Fann

REFERENCES:
- [Derived] Benzekri NA, Sambou JF, Tamba IT, Diatta JP, Sall I, Cisse O, Thiam M, Bassene G, Badji NM, Faye K, Sall F, Malomar JJ, Seydi M, Gottlieb GS. Nutrition support for HIV-TB co-infected adults in Senegal, West Africa: A randomized pilot implementation study. PLoS One. 2019 Jul 18;14(7):e0219118. doi: 10.1371/journal.pone.0219118. eCollection 2019. PMID 31318879